CLINICAL TRIAL: NCT06310109
Title: Effect of Pediatric Intensive Care Unit (PICU) Diaries on the Post Intensive Care Syndrome (PICS-p) in Children and Young Adults and Their Caregivers
Brief Title: Effect of Pediatric Intensive Care Unit Diaries on PICS-p
Acronym: PICS-p
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Children's Hospital IRCCS (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Orsola Gawronski, Principal Investigator, Bambino Gesù Children's Hospital IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2358_OPBG 2020
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Post Intensive Care Syndrome; Narrative Medicine; Post Traumatic Stress Disorder; Anxiety; Depression
Keywords: Post Intensive Care Syndrome; Pediatric; Children; Diary; ICU diary; Narrative medicine; Pediatric Intensive Care Unit
MeSH Terms: conditions — postintensive care syndrome; Narrative Medicine; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICU diary (Experimental): The "PICU diary" arm, will receive a PICU diary at the patient bedside.
  Interventions: Other: PICU diary
- Control arm (No Intervention): The control arm will receive standard care (no PICU diary).

INTERVENTIONS:
Other: PICU diary — .The PICU diary is a notebook with lined sheets located at the patient's bedside. In this diary parents, other caregivers, family members, healthcare professionals or other visitors can write thoughts, report events related to the child/adolescent's admission, attach drawings or photographs for the patient or related to the PICU admission.
  Other Names: Journal
  Arms: PICU diary

SUMMARY:
When children become very sick and need to stay in a Pediatric Intensive Care Unit (PICU), it can have a big impact on their recovery and their family's well-being. Sometimes kids and their families feel worried or sad even after they leave the hospital. This can have an impact on the quality of their life after hospital discharge.

To help understand and improve these experiences, the investigators want to study the "PICU diaries." These are journals that families and hospital staff can write in during the child's time in the hospital. Parents, other visitors and healthcare professionals can share thoughts, experiences, and even drawings or photos related to the child's admission. The content is a narrative account of what happens during the child's hospital stay, for the family to take home at PICU discharge.

The investigators believe that writing in these diaries might help children and their families feel better after leaving the hospital. It might help kids feel less worried or sad, and it might also help their parents or caregivers feel better too.

The study will include children who have been in the PICU and their families. Some families will receive these special diaries to use during their time in the hospital, while others won't. We'll then see how everyone feels after they leave the hospital and compare the two groups to see if the diaries make a difference.

The investigators hope that by understanding how these diaries can help, healthcare professionals can make hospital experiences better for everyone involved.

ELIGIBILITY:
Inclusion Criteria:

* children/adolescents admitted to the PICU
* Mechanical ventilation for > 48 hours
* Patient's age <19 years old

Exclusion Criteria:

* parents who are unable to communicate in Italian language
* parents who have not signed and informed consent
* patients with a poor prognosis

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Parent's Post Traumatic Stress Disease (PTSD) | Through study completion, an average of 3 year
  The PTSD Checklist according to the Diagnostic and Statistical Manual of Mental Disorders (PCL-5) will be used to measure parent's post traumatic stress after PICU discharge.
Parent's Anxiety | Through study completion, an average of 3 year
  The Generalized Anxiety Disorder - 7 scale (GAD-7) will be used to measure parent's anxiety.
Child's Strengths and difficulties | Through study completion, an average of 3 year
  The Strengths and Difficulties Questionnaire (SDQ), a brief behavioural screening questionnaire about 2-17 year olds wukk be used.
Child's Post Traumatic Stress Disease (PTSD) | Through study completion, an average of 3 year
  The child's PTSD will be measured using the Revised Child Impact of Event Scale - (R CRIES 8)
Child's Anxiety | Through study completion, an average of 3 year
  The Generalized Anxiety Disorder - 7 scale (GAD-7) will be used to measure the child's anxiety disorder.
Child's Depression | Through study completion, an average of 3 year
  The Patient Health Questionnaire-9 (PHQ-9) will be used to measure the child's depression.

SECONDARY OUTCOMES:
Satisfaction with PICU care | Through study completion, an average of 3 year
  Satisfaction with PICU care will be measured using The EMpowerment of PArents in The Intensive Care (EMPATHIC-P).
Patient's Quality of Life | Through study completion, an average of 3 year
  The Quality of Life will be measured using the Pediatric Quality of Life Inventory (PedsQL).

CONTACTS AND LOCATIONS:
Overall Officials: Orsola Gawronski, PhD, Principal Investigator — Bambino Gesù Children's Hospital IRCCS
Locations (1):
- Bambino Gesù Children's Hospital IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No
Limited dataset, pilot study.